CLINICAL TRIAL: NCT00714428
Title: Development of a Quality of Life Tool for Deployment Related TBI
Brief Title: Development of Quality of Life Tool for TBI
Acronym: TBIQOL
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: Northwestern University (Other); University of Michigan (Other)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: B6237-R
Record Dates: First submitted 2008-07-08; First posted 2008-07-14 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Quality of Life
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — None retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1: Item Development: Individuals with TBI to provide input to relevant questions for quality of life measure in TBI
- Group 2: Item Development: Clinicians who treat those with deployment related TBI to obtain their feedback on relevant questions pertaining to quality of life measures in TBI.
- Group 3: Instrument Development: Individuals with deployment TBI who will complete the Beta version of the TBI QOL measure.

SUMMARY:
Objectives: The ultimate goal of this research program is to promote seamless, comprehensive care for Operation Enduring Freedom/ Operation Iraqi Freedom (OEF/OIF) veterans. The purpose of this study is to develop a psychometrically sound tool to measure health-related quality of life (HRQOL) applicable to wounded warriors with TBI (deployment-related TBI).

DETAILED DESCRIPTION:
Specific short-term objectives for this study include:

O1: Identify a parsimonious set of domains that capture HRQOL in deployment-related TBI.

O2: Construct and refine clinically-relevant HRQOL of life item banks for deployment-related TBI, in order to supplement the TBI-QOL and generic Neuro-QOL banks and extend the TBI/Neuro-QOL projects to address the unique issues facing wounded warriors with TBI.

O3:Utilize Item Response Theory methodology to refine and calibrate targeted and generic item banks for use with deployment-related TBI.

O4:Develop a short form, refining item sets and developing algorithms for future development of a computerized adaptive test.

Research Design: The proposed three-year prospective study will employ a mixed methods research design in three stages. Combining qualitative and quantitative methods maximizes the ability of the study team to design and validate a clinically sensitive HRQOL measure for wounded warriors with deployment-related TBI. Furthermore, this approach is consistent with the FDA's draft guidance on patient reported outcome (PRO) measures development.

Phase 1: Qualitative data obtained from focus groups of veterans and VA providers will be used to (a) evaluate the generic Neuro-QOL domains and items for relevance and appropriateness for use in deployment-related TBI and (b) identify new HRQOL domains and items specific to deployment-related TBI. [Objective #1] Phase 2: The generic and specific item banks will be field tested in a large sample of veterans with deployment-related TBI recruited from all 4 VA Polytrauma Rehabilitation Centers (PRCs). [Objective #2] Phase 3: Psychometric analyses, including item response theory (IRT) of field test data will be completed. The psychometric properties of the scale will be evaluated empirically. A short form will be developed, refining item sets and developing algorithms for future development of a computerized adaptive test (CAT). [Objectives #3 & 4]

ELIGIBILITY:
Inclusion Criteria:

* enrolled in VA and diagnosed with a deployment-related TBI documented in computerized patient record system (CPRS)
* at least one year post injury
* greater than 18 years of age
* able to follow two step commands and
* English speaking

Clinicians Inclusion Criteria:

* Clinicians, including:

  * physicians
  * psychologists
  * nurses
  * social workers
  * therapists who have provided care to wounded warriors with deployment-related TBI for at least three years

Exclusion Criteria:

Veterans Exclusion criteria include:

* those veterans who are not yet discharged from initial rehabilitation (want patients to experience community based living environment)
* living in the community less than three months post initial rehabilitation, including residential care or long term care living environments

No exclusion criteria for the clinicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with deployment related traumatic brain injury and clinicians who treat those veterans.
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2009-04; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
development of an outcomes measure | one time

CONTACTS AND LOCATIONS:
Overall Officials: Rodney D Vanderploeg, PhD, Principal Investigator — James A. Haley Veterans' Hospital
Locations (4):
- United States (4):
  - VA Palo Alto Health Care System, Palo Alto, California
  - James A. Haley Veterans' Hospital, Tampa, Florida
  - VA Medical Center, Minneapolis, Minneapolis, Minnesota
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia

REFERENCES:
- [Result] Toyinbo PA, Vanderploeg RD, Donnell AJ, Mutolo SA, Cook KF, Kisala PA, Tulsky DS. Development and Initial Validation of Military Deployment-Related TBI Quality-of-Life Item Banks. J Head Trauma Rehabil. 2016 Jan-Feb;31(1):52-61. doi: 10.1097/HTR.0000000000000089. PMID 25310294